CLINICAL TRIAL: NCT01393548
Title: Multicenter, Phase III, Randomized, Open, Parallel, Comparative to Evaluate the Efficacy and Safety of the Treatment of Nasal Congestion and Runny Nose Present in Acute Crisis of Viral Rhinitis and Allergic Reactions, in Pediatric Patients
Brief Title: Efficacy and Safety of Combination of Brompheniramine and Phenylephrine for the Symptoms Relief of Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-DCN-03(03/10)
Record Dates: First submitted 2010-10-27; First posted 2011-07-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Nasal Congestion and Inflammations; Rhinitis
Keywords: Rhinitis; common cold; nasal symptoms; children
MeSH Terms: conditions — Nasal Obstruction; Inflammation; Rhinitis; Common Cold | interventions — brompheniramine, pseudoephedrine drug combination; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- brompheniramine + phenylephrine (Experimental): Fixed dose combination of brompheniramine + phenylephrine
  Interventions: Drug: brompheniramine + phenylephrine
- brompheniramine + pseudoephedrine (Active Comparator): Fixed dose combination of brompheniramine + pseudoephedrine
  Interventions: Drug: Brompheniramine + pseudoephedrine

INTERVENTIONS:
Drug: brompheniramine + phenylephrine — Oral solution: brompheniramine (2mg/mL) and phenylephrine (2,5 mg/mL), t.i.d., according weight of patient.
  OR Syrup: brompheniramine (2mg/5mL) and phenylephrine(5 mg/5mL), t.i.d., according weight of patient.
  Other Names: Group 1
  Arms: brompheniramine + phenylephrine
Drug: Brompheniramine + pseudoephedrine — Elixir: Brompheniramine (0,2mg/mL) and pseudoephedrine (3,0 mg/mL), t.i.d., according weight of patient
  Other Names: Group 2
  Arms: brompheniramine + pseudoephedrine

SUMMARY:
This is a multicenter clinical trial, phase III, non-inferiority, controlled by active medicine, open, randomized, enroll 538 children, 2 to 12 years old, with acute inflammation upper airway, characterized by nasal congestion and runny nose, lasting at least 24 hours and a maximum of 48 hours prior to inclusion. The subjects will be allocated in 2 parallel groups, and will receive the medicines of study, according of the randomization.

DETAILED DESCRIPTION:
This study evaluate the efficacy and safety of experimental drug The study was designed to evaluate the efficacy and safety of fixed combinations Decongex® Plus Syrup and Decongex® Plus Oral Solution (consisting of brompheniramine maleate and phenylephrine hydrochloride) compared to Resfenol® Oral Solution (paracetamol, maleate chlorpheniramine and phenylephrine hydrochloride) in the treatment of nasal congestion and rhinorrhea present in acute attacks of viral rhinitis (common cold) and allergic. This study population will consist in participants of both sexes, aged between 6 to 11 years old with acute inflammatory condition of the upper airways, defined as nasal congestion and runny nose, with no less than 24 (twenty four) hours and a maximum of 48 (forty-eight) hours prior to inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 2 and 12 years old, of both sexes. Must be responsible be able to understand and provide ICF and able to allow compliance to treatment and protocol requirements, fulfilling the regular visits;
2. Patients with symptoms of acute inflammation upper airway, starting between 24 and 48 hours of their inclusion in this study protocol;
3. Presence of runny nose classification moderate or severe (score 2 or 3), according the responsible evaluation;
4. Presence of nasal congestion classification moderate or severe (score 2 or 3), according the responsible evaluation.

Exclusion Criteria:

1. Patients younger than 2 years or percentile for body weight and/or height less than 25;
2. History of nasal obstruction in chronic rhinosinusitis and / or nasal polyposis;
3. Oral chronic respirator with history for six months;
4. Personal history of nasal surgery that in the opinion of the investigator can influence the resistance to nasal airflow;
5. Patients who have a clinical history confirmed (diagnosed) with asthma;
6. Patients under medicine treatment for chronic allergy;
7. Patients with gastroesophageal reflux disease;
8. Presence of psychiatric illness of any kind;
9. Presence of mental retardation from any cause;
10. Diagnosis of renal or hepatic failure;
11. Patients with genetic syndromes;
12. History of hypersensitivity to (s) drug (s) of study or their excipients;
13. Use of prohibited medicine within the prescribed period before the V0 - Inclusion Visit (Table 1);
14. Patients who participated in the last 12 months, of clinical trials protocols;
15. Patients who didn´t updated vaccine book;
16. Relatives of sponsor´s or study site´s employee;
17. Suggestive signs of bacterial infection of upper airways at rhinoscopy, otoscopy or oroscopy;
18. Presence of anemic/inflamed turbinate at anterior rhinoscopy;
19. Presence of septal deviation grade II and III (in any region and any nasal cavity) and / or nasal polyps, or other conditions determinants of nasal obstruction;
20. Presence of purulent or mucopurulent secretion, nasal vault or mal formations (cleft lip or cleft nasolabial corrected or not) in nasal vestibule;
21. Current evidence of clinically significant diseases: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrine, psychiatric, autoimmune, pulmonary, or another disease that block the patient participation;
22. Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the patient or interfere with the endpoints of study.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 879 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement of nasal congestion and runny nose, after 48 hours of treatment | 48 hours after single dose of double-blind treatment
  Improvement is defined as a reduction of at least one point on the rating scale, in both nasal symptoms, after 48 hours of treatment.
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.

SECONDARY OUTCOMES:
Overall score of nasal and extranasal symptoms (nasal congestion, runny nose, sneezing, watery eyes and itching) | After 2 and 5 (± 1) days of treatment
Clinical score of upper airway compromise | After 2 and 5 (± 1) days of treatment
Proportion of subjects who used at least once the rescue medication | Within 2 days and the period of 5 (± 1) days of treatment
Safety descriptive about occurence of adverse events, evaluation of results of general physical examination. | Will be evaluated during the 5(± 1) days of treatment
  Collection of safety data throughout the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Fábio M Castro, Principal Investigator — IMA
Locations (1):
- Ache Laboratorios Farmaceuticos, Guarulhos, São Paulo, Brazil